CLINICAL TRIAL: NCT04844502
Title: Cardiopulmonary Function and Quality of Life in People With Sequelae of Pulmonary Tuberculosis Undergoing Pulmonary Rehabilitation: Controlled and Randomized Study.
Brief Title: Cardiopulmonary Function and Quality of Life in Pulmonary Tuberculosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Diego de Faria Magalhães Torres, Diego de Faria Magalhães Torres, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10481219.9.0000.5257
Record Dates: First submitted 2021-04-10; First posted 2021-04-14 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Tuberculosis, Pulmonary; Physical Disability; Quality of Life
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Frequent life activities.
- Intervention Group (Experimental): Protocol of physical exercises
  Interventions: Other: Physical rehabilitation

INTERVENTIONS:
Other: Physical rehabilitation — Rehabilitation can be applied to the intervention group in two ways: in person or by home orientation. The face-to-face form will correspond to 5 weeks of intervention, 3 sessions per week, which should include: a) aerobic resistance training of 30 minutes in total, five minutes of cooling down); b) strengthening of peripheral muscles using 20-minute sessions of calisthenic exercises; and c) maintained active stretching, for 10 minutes, for the main muscle groups. The home-based intervention will correspond to three months of daily activities, monitored twice a week in the first month and once a week in the second and third months, by telephone or video conference, and will follow an exercise protocol that includes: a) aerobic resistance training for 15 uninterrupted minutes; b) anaerobic training to strengthen the peripheral muscles for 15 minutes at intervals with breathing exercises; and c) maintained active stretching, for 10 minutes, for the main muscle groups.
  Arms: Intervention Group

SUMMARY:
This work aims to assess cardiopulmonary function and quality of life in people with sequelae of pulmonary tuberculosis undergoing rehabilitation. It is an experimental clinical study, with evaluation before and after the intervention. Included participants will be randomized and divided into a control group and an intervention group. Quality of life is examined by two questionnaires and physical fitness by specific tests, before and after the intervention. The intervention is the realization of a supervised physical exercise protocol.

DETAILED DESCRIPTION:
Experimental clinical study, with evaluation before and after intervention, for a determined period of two years for data collection and one year for analysis and publication of results. Included participants will be randomized and divided into a control group and an intervention group.

People with sequelae of pulmonary tuberculosis undergoing follow-up at the pulmonology outpatient clinic will be invited to participate in this study, with an estimated sample of 60 participants, according to the following criteria:

1. Inclusion: people diagnosed with treated pulmonary tuberculosis, with negative culture in induced sputum; with pulmonary function report (spirometry), chest X-ray and complete blood count with biochemistry updated in the last month, and in accordance with the Informed Consent Form.
2. Exclusion: people with non-cooperative pulmonary tuberculosis, who present clinical instability and / or musculoskeletal injury that compromises pulmonary rehabilitation and limits the perception of physical capacity; with any comorbidities that may cause or accentuate dyspnea; with stable angina, severe arrhythmias and / or heart failure.

Protocols:

1. Anamnesis and medical record examination

   The anamnesis and examination of the medical records of the research participants will be carried out through outpatient scheduling for adequate availability of the medical records, by the main researcher. The evaluation will consist of searching for the following main information: a) complaint and history of the disease; b) time of diagnosis of pulmonary tuberculosis; c) medications used in the treatment; d) duration of use of medications for treatment; e) age of the participant; and f) gender of the participant.
2. Physical examination

   The physical examination will consist of the analysis of the following data and respective instruments and collection procedures: a) Anthropometry - the bioimpedance equipment by tetrapolar technique (InBody 230® Bioscope - Seoul - Korea) will be used, with bare feet, with light clothing and will consist of the verification of the following data: body mass, body height and Body Mass Index (BMI); b) Systemic blood pressure - measured using an aneroid sphygmomanometer, analog with a smaller division of 2 mmHg, Brand: Premium® (certified by INMETRO), applied to the left arm, associated with the auscultatory method for determining systolic systemic blood pressure (SBP) and systemic diastolic blood pressure (SBP); c) Partial oxygen saturation - measured using a portable pulse oximeter (model 9500; Nonin Medical Inc., Minneapolis, USA), with a sensor positioned on the 2nd finger of the right hand, the reading being determined after signal stabilization, obtaining the partial arterial percentage of saturated oxygen (SpO2); d) Heart rate (HR) - measured using a portable pulse oximeter (model 9500; Nonin Medical Inc., Minneapolis, MN, USA), applied to the index finger of the left hand, obtaining the number of heart beats in one minute (bpm); e) Respiratory frequency (RF) - measured by counting by observing the thoracoabdominal movement of the number of respiratory incursions in one minute (irpm); f) Pulmonary auscultation - verification of lung sounds using a stethoscope; g) Cardiac auscultation - verification of cardiac sounds through the use of a stethoscope.
3. Complementary exams

   They comprise routine examinations performed on these participants during the phase preceding the research, for diagnosis and clinical treatment, therefore inserted only as procedures for analysis of the reports and classification.

   Simple chest X-rays, lateral and postero-anterior views, corresponding to the last month of clinical treatment and submitted to the classification of the National Tuberculosis Association (NTA) will be analyzed.

   The pulmonary function tests or spirometry will be analyzed in accordance with the Guidelines for Pulmonary Function Tests of the Brazilian Society of Pulmonology.

   The analysis of the complete blood count and blood biochemistry will consist of the observation between the normal values of the following items: hematocrit, total leukocytes, neutrophils, eosinophils, lipogram, glucose, glycated hemoglobin, albumin, urea, creatinine, liver enzymes and C reactive protein.
4. Examination of mental status

   The Mini Mental State Examination (Mini-mental) will be applied, a test that allows a quick and objective assessment of the research participant's cognitive function.
5. Quality of life assessment

   The Questionnaire of the Hospital Saint George on Respiratory Illness (SGRQ) will be applied, specific for assessing the quality of life in respiratory diseases that addresses the impacts of the disease on individuals in three areas or domains: symptoms, activity and psychosocial aspects. Another instrument used to assess quality of life is the Short-Form 36 (SF-36), a generic questionnaire, self-administered or applied by interview, consisting of 36 items that assess the domains: functional capacity, physical aspects, pain, condition general health, vitality, social aspects, emotional aspects and mental health.
6. Functional assessment

   The perception of effort will be measured by presenting the Modified Dyspnea Scale (Borg). The Medical Research Council Classification for dyspnoea will also be applied.

   For the assessment of disabilities in instrumental activities of daily living (IADLs), the scale developed by Lawton and Brody (1969) will be applied. The frailty assessment will also be carried out on the research participants through the clinical frailty scale.
7. Physical evaluation

The six-minute walk test will be performed, a submaximal test used to assess the distance covered by the participant in six uninterrupted minutes, with monitoring of blood pressure, heart rate (HR), modified BORG scale and oxygen saturation (SpO2), in a 50-meter, flat corridor, with demarcated distances meter by meter, following the recommendations of the American Thoracic Society. The sit and stand test will also be applied five times, a functional test that reproduces an everyday activity that particularly depends on the strength of the muscles of the lower limbs and body balance.

Static spirometry test will be applied to assess respiratory muscle strength. This method is performed by measuring the Maximum Inspiratory Pressure (MIP) and Maximum Expiratory Pressure (MEP).

To assess peripheral muscle strength, isokinetic dynamometry of the lower limbs will be used. The equipment used will be the Biodex System® dynamometer. The participant will adopt the sitting posture on the device with an inclination of +/- 100 degrees (internal angle), with the motor axis aligned with the knee joint axis and stabilizations in the trunk, hip and thigh to avoid compensations related to the maximum effort. The lever arm will be positioned at the distal third of the tested leg (three centimeters proximal to the tibial malleolus). The execution speeds to be tested for quadriceps and hamstrings will be 75º / s and 240º / s (4 repetitions), in amplitudes of 100º - 0º, with a resting time of two minutes.

Reassessments will be made after one, three and six months of intervention.

Intervention protocol:

Rehabilitation can be applied to the intervention group in two ways: in person or by home orientation. The face-to-face form will correspond to 5 weeks of intervention, 3 sessions per week, which should include: a) aerobic resistance training (performed with a bicycle or treadmill) of 30 minutes in total (five minutes of warm-up, 20 minutes of aerobic training) , five minutes of cooling down); b) strengthening of peripheral muscles using 20-minute sessions of calisthenic exercises; and c) maintained active stretching (stretching), for 10 minutes, for the main muscle groups. The minimum adherence to the training sessions is 80% and all sessions will be accompanied by a doctor from the institution for effective first aid if necessary.

The home orientation intervention (telerehabilitation) will correspond to three months of daily activities, monitored twice a week in the first month and once a week in the second and third months, by telephone or video conference, and will follow an exercise protocol that includes: a) aerobic resistance training (walking, cycling, swimming or step exercises) for 15 uninterrupted minutes; b) anaerobic training to strengthen the peripheral muscles (calisthenic exercises) for 15 minutes at intervals with breathing exercises; and c) maintained active stretching (stretching), for 10 minutes, for the main muscle groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Pulmonary Tuberculosis,
* negative culture in induced sputum;
* pulmonary function report (spirometry), chest X-ray and complete blood count with biochemistry updated in the last month,
* in accordance with the Informed Consent Form.

Exclusion Criteria:

* Non-cooperative patients,
* clinical instability and / or musculoskeletal injury that compromises Pulmonary Rehabilitation and limits the perception of physical capacity;
* comorbidities that may cause or accentuate dyspnea (Asthma, COPD, Pulmonary Fibrosis, Obesity);
* stable angina, severe arrhythmias and / or heart failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Physical Capacity | 9 months
  Comparison between a physical capacity evaluation

SECONDARY OUTCOMES:
Quality of Life reported | 9 months
  Comparison between a quality of life evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No